CLINICAL TRIAL: NCT06155240
Title: Yoga for a Healthy Heart Study: Addressing Stress Management and Functional Cognition as Barriers to Both Medication Management and Blood Pressure Regulation for African American Patients With Hypertension
Brief Title: Yoga for a Healthy Heart
Acronym: YHH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Allan Chiunda, Principle Investigator, The Brentwood Foundation Chair in Research and Data Analytics | Director of Cleveland Clinic South Pointe Hospital Clinical Effectiveness, Initiatives and Innovations, MD, PhD, MPH, The Cleveland Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-445
Record Dates: First submitted 2023-11-02; First posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Single cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Yoga participant (Experimental): Providing once weekly class for 8 weeks, participants will take part in performing yoga poses and yoga breathing and meditation for stress management
  Interventions: Behavioral: Therapeutic yoga

INTERVENTIONS:
Behavioral: Therapeutic yoga — Yoga interventions include yoga poses, breathing, and meditation

SUMMARY:
The Yoga for a Healthy Heart study will address various barriers to both medication management and blood pressure regulation for African American patients with hypertension.

DETAILED DESCRIPTION:
The program will take place in person at South Pointe's hospital community outreach center. The program will be an 8-week program, once per week, 60 minutes in length, consisting of meditation, or relaxation, pranayama which are breathing techniques and asana, or physical postures. Yoga, is defined as the fluctuations or roaming tendencies of the mind according the Patanjali's Yoga Sutras. In addition to therapeutic yoga techniques, lifestyle management will be discussed or self-reflections written in journals. Lifestyle management skills include learning how to take blood pressure and manage a pillbox, as well as develop prosocial communication skills through lessons on mindful communication. The classes will be taught in person. The instructor facilitating the program will be a skilled healthcare professional certified in both Occupational Therapy and Yoga teaching at the 500-hour level. The Occupational Therapist will provide both skilled assessments and interventions in the group setting of the community health class. Assessments include: 1. Perceived Stress Scale 2. Canadian Occupational Performance Measurement 3. Mini and Medi-Cog 4. Blood pressure assessments pre and post class.

.

ELIGIBILITY:
Inclusion Criteria:

* Over 18
* has transportation to South Pointe Hospital
* Has the ability to walk, or use a wheelchair from the entrance of the building
* Able to attend all 8 sessions
* Diagnosis of hypertension
* African American
* Prescribed antihypertensive medication
* Able to stand up from the chair independently
* Able to walk to the bathroom independently with or without a device
* Approved by cardiologist to participate

Exclusion Criteria:

* Unable to tolerate sitting for 1 hour
* BP over 200/100
* Unable to independently walk or use a wheelchair to the bathroom

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2024-05-11 (Estimated); Study Completion 2024-05-11 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | 8 weeks
  take both systolic and diastolic blood pressure before and after intervention each class and from beginning of session to end of 8 week session
Perceived Stress Scale (PSS) | 8 weeks
  Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress. Scores ranging from 27-40 would be considered high perceived stress. To assess changes in outcomes for perceived stress from beginning of intervention to completion of intervention
Canadian Occupational Performance Measurement | 8 weeks
  Changes in components of the COPM that reflect self-care, productivity, and leisure activities may also be analyzed separately in a similar manner using the participants that have rated a problem within these categories among the 5 most important problems used to calculate their total COPM score.
Mini and Medi Cog | 8 weeks
  To assess changes in outcomes on managing medications and on short term memory

CONTACTS AND LOCATIONS:
Overall Officials: Allan Chiunda, MD, PhD, Principal Investigator — South Pointe Hospital
Locations (1):
- South Pointe Hospital, Warrensville Heights, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aggarwal M, Bozkurt B, Panjrath G, Aggarwal B, Ostfeld RJ, Barnard ND, Gaggin H, Freeman AM, Allen K, Madan S, Massera D, Litwin SE; American College of Cardiology's Nutrition and Lifestyle Committee of the Prevention of Cardiovascular Disease Council. Lifestyle Modifications for Preventing and Treating Heart Failure. J Am Coll Cardiol. 2018 Nov 6;72(19):2391-2405. doi: 10.1016/j.jacc.2018.08.2160. PMID 30384895
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Ferdinand KC, Yadav K, Nasser SA, Clayton-Jeter HD, Lewin J, Cryer DR, Senatore FF. Disparities in hypertension and cardiovascular disease in blacks: The critical role of medication adherence. J Clin Hypertens (Greenwich). 2017 Oct;19(10):1015-1024. doi: 10.1111/jch.13089. Epub 2017 Aug 30. PMID 28856834
- [Background] Lam AY, Anderson K, Borson S, Smith FL. A pilot study to assess cognition and pillbox fill accuracy by community-dwelling older adults. Consult Pharm. 2011 Apr;26(4):256-63. doi: 10.4140/TCP.n.2011.256. PMID 21486736
- [Background] Lorig KR, Sobel DS, Stewart AL, Brown BW Jr, Bandura A, Ritter P, Gonzalez VM, Laurent DD, Holman HR. Evidence suggesting that a chronic disease self-management program can improve health status while reducing hospitalization: a randomized trial. Med Care. 1999 Jan;37(1):5-14. doi: 10.1097/00005650-199901000-00003. PMID 10413387
- [Background] Beech BM, Ford C, Thorpe RJ Jr, Bruce MA, Norris KC. Poverty, Racism, and the Public Health Crisis in America. Front Public Health. 2021 Sep 6;9:699049. doi: 10.3389/fpubh.2021.699049. eCollection 2021. PMID 34552904
- [Background] Basu-Ray I, Mehta DH, Shah S. Initial Treatment of Hypertension. N Engl J Med. 2018 May 17;378(20):1952-3. doi: 10.1056/NEJMc1804084. No abstract available. PMID 29770683
- [Background] Pullen PR, Thompson WR, Benardot D, Brandon LJ, Mehta PK, Rifai L, Vadnais DS, Parrott JM, Khan BV. Benefits of yoga for African American heart failure patients. Med Sci Sports Exerc. 2010 Apr;42(4):651-7. doi: 10.1249/MSS.0b013e3181bf24c4. PMID 19952833
- [Background] Rana J, Oldroyd J, Islam MM, Tarazona-Meza CE, Islam RM. Prevalence of hypertension and controlled hypertension among United States adults: Evidence from NHANES 2017-18 survey. Int J Cardiol Hypertens. 2020 Oct 26;7:100061. doi: 10.1016/j.ijchy.2020.100061. eCollection 2020 Dec. PMID 33447782
- [Background] Sorrentino MJ. The Evolution from Hypertension to Heart Failure. Heart Fail Clin. 2019 Oct;15(4):447-453. doi: 10.1016/j.hfc.2019.06.005. Epub 2019 Aug 7. PMID 31472880
- [Background] Ziaeian B, Fonarow GC. The Prevention of Hospital Readmissions in Heart Failure. Prog Cardiovasc Dis. 2016 Jan-Feb;58(4):379-85. doi: 10.1016/j.pcad.2015.09.004. Epub 2015 Oct 21. PMID 26432556

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-06): https://cdn.clinicaltrials.gov/large-docs/40/NCT06155240/Prot_SAP_000.pdf